CLINICAL TRIAL: NCT04731961
Title: Reduced Site Injection Protocol of Intra-detrusor Onabotulinumtoxin-A for Treatment of Idiopathic Refractory Urgency Urinary Incontinence
Brief Title: Reduction in Number of Botox Injections for Urgency Urinary Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Monique Vaughan, MD, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSR200175
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Urgency Urinary Incontinence
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to arms with either 5 or 15 injections.
Who Masked: Participant
Masking Description: The patients will not be informed of which arm they are assigned to before the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Controls (Active Comparator): Subjects in this arm will be administered the standard injection site protocol (15 sites).
  Interventions: Procedure: Standard of care (15 Botox injections)
- Experimental (Experimental): Subjects in this arm will be administered the same amount of Botox in 5 injection sites.
  Interventions: Procedure: Experimental Arm (5 Botox injections)

INTERVENTIONS:
Procedure: Standard of care (15 Botox injections) — The controls will be given the standard of care of 15 Botox injections.
  Arms: Controls
Procedure: Experimental Arm (5 Botox injections) — 5 Botox injections will be given, with each injection containing three times the amount of Botox than each of the 15 injections given in the standard of care arm.
  Arms: Experimental

SUMMARY:
The overall objective of this study is to determine if a reduced injection site protocol (5 injection sites) using an equivalent amount of Botox provides comparable relief of Urgency Urinary Incontinence (UUI) symptoms compared to the standard injection site protocol (15-20 injection sites). Our central hypothesis is that the 5-site injection protocol is non-inferior in terms of relief of UUI symptoms compared to the standard injection site protocol, measured by a non-inferior reduction in the number of UUI episodes per day.

DETAILED DESCRIPTION:
English speaking women ≥21 years old with idiopathic refractory urgency urinary incontinence who have failed first and second line treatment (life style modifications and antispasmodic medications) who are undergoing a first injection of intra-detrusor Botox will be recruited to participate in this study. Failure of first and second line treatment will be defined as no improvement in urgency urinary incontinence episodes after trial of lifestyle modifications and use of at least one antispasmodic agent.

Patients who are planning to undergo her first intra-detrusor Botox procedure for refractory idiopathic urgency urinary incontinence at the University of Virginia Pelvic Medicine and Reconstructive Surgery clinic will be approached for inclusion into the study. A study overview, as well as risks and benefits, will be reviewed with the patients. The patient will be screened for inclusion/exclusion criteria. If she meets criteria and agrees to study participation, she will be consented for study participation and the Botox injection procedure.

Prior to receiving treatment, patients will complete a 3-day voiding diary and the following questionnaires: Incontinence Impact Questionnaire short form (IIQ-7) and Urogenital Distress Inventory short form (UDI-6) at the time of consent. As part of usual care, patients in both arms will receive prophylactic antibiotics (oral nitrofurantoin or cephalexin) to complete prior to the procedure date. On the day of treatment, patients will have a clean catch urine specimen obtained and urine dip completed. Patients who have a positive urine dip will have her procedure rescheduled to another day. A positive urine dip is defined as + leukocytes and + blood in the presence of symptoms of urinary tract infection (dysuria, increased urgency/frequency above baseline or hematuria). In this study, we will not offer patients pre-procedure oral Valium as it may affect reporting of pain scores. Patients in both arms will be prepared for the procedure in the same fashion: 50 cc of 1% lidocaine will be instilled into the bladder at least 20 minutes prior to the procedure. Patients will then be prepped and draped in the standard fashion. A 70-degree cystoscope will be inserted through the urethra and into the bladder until the trigone is identified; the bladder will be distended with approximately 200 mL sterile saline.

100 units of Botox will be mixed with 10 mL of Normal Saline for sterile injection into the bladder. In the reduced protocol arm, a single row of 5 injections will be administered into the detrusor muscle. In the standard protocol arm, 3 rows of 5 injections will be administered into the detrusor muscle. In both arms, a final injection with 1 mL of normal saline flush will be injected to remove any residual Botox from the injection needle. The patient will be monitored for 20 minutes post procedure to ensure adequate ability to void after treatment. Approximately 5 minutes post-procedure, patients will rate their pain experienced during the procedure using a 100-point visual analog pain scale.

If the patient is unable to void post-procedure, she will be taught how to perform clean intermittent self-catheterization (CISC) and provided with a log to record void and catheter volumes. She will be called on a weekly basis by the study team to review void/catheterization volumes and encouraged to discontinue when she has 2 successive catheterization volumes of <150 ml. This is in accordance with standard clinical care in our practice.

At 2 weeks post procedure, patients in both treatment arms will be interviewed by phone to report results of a 3-day voiding diary (Aim 1), complete the IIQ-7 and UDI-6 again, as well as the OAB Treatment Satisfaction Questionnaire (OAB-SATq), Client Satisfaction Questionnaire (CSQ-8)10, Patient Global Impression of Improvement (PGI-I) questionnaire and evaluate for complications (Aim 2, Aim 3). The same evaluation process will be repeated at 3 months and 6 months post procedure.

After completion of all questionnaires at the 4 timepoints (Pre-procedure, 2 weeks, 3 months, 6 months), patients will receive a $50 incentive for their time and participation.

ELIGIBILITY:
Inclusion Criteria:

* Females at least 21 years of age
* English speaking
* Five or more urge urinary incontinence episodes on a three-day voiding diary. Urge incontinence episodes will be determined based on voiding diary and subject indication of coincident urge symptoms, allowing for self-characterization of incontinence type
* Urge predominant (urge >50% of total incontinent episodes) urinary incontinence based on self-reported characterization of incontinent episodes on diary
* Patient or caregiver willing to perform clean intermittent catheterization, or patient willing to have indwelling Foley catheter in the event this would be required
* Request for treatment for urgency urinary incontinence. The patient may have tried other pharmacologic treatments for urge incontinence, such as antispasmodic agents or non-pharmacologic treatments, such as supervised behavioral therapy, supervised physical therapy, unsupervised physical therapy, supervised biofeedback, and transvaginal electrical stimulation.
* Subject has undergone 3-week washout period if subject were on anticholinergic therapy prior to enrollment
* Subject is able to complete all study related items and interviews
* Willingness and ability to comply with scheduled visits and study procedures.

Exclusion Criteria:

* Current symptomatic urinary tract infection that has not resolved prior to randomization.
* Baseline need for intermittent self-catheterization
* PVR (Post void residual) >150 mL on 2 occasions with void(s) of greater than 150 mL
* Surgical treatment for stress incontinence (sling, Burch or urethral injection) or pelvic organ prolapse recommended or planned at enrollment by study investigator(s).
* Any prior intra-detrusor botulinum toxin A injections
* Previous or currently implanted neuromodulation (sacral or tibial).
* Surgically altered detrusor muscle, such as augmentation cystoplasty.
* Known allergy to botulinum toxin A.
* Women with known neurologic disease believed to potentially affect urinary function (history of stroke, Parkinson's disease, multiple sclerosis, spinal cord injuries, myasthenia gravis, Charcot-Marie-Tooth disease).
* Known allergy to lidocaine.
* Currently pregnant or lactating patients or patients planning pregnancy within the next year.
* Sexually active premenopausal women with a uterus who have either not had a tubal ligation or are not on a medically approved form of contraception for at least 3 months prior to and throughout the duration of the study.
* Cystoscopic findings that preclude injection, in the opinion of the investigator.
* Current or prior bladder malignancy.
* Inability to understand diary instructions and complete 3-day voiding diary.
* Subject has been previously diagnosed with interstitial cystitis or chronic pelvic pain syndrome.
* Subjects with hematuria who have not undergone a clinically appropriate evaluation.
* Serum creatinine level greater than twice the upper limit of normal within the previous year.
* Two or more hospitalizations for medical conditions in the previous years
* Plans to move out of area in the next 6 months

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Reducton of Urgency Urinary Incontinence episodes in standard of care versus modified treatment group | 6 months
  To determine if a reduced injection site protocol (5 injection sites) of intra-detrusor Onabotulinumtoxin-A is non-inferior in the treatment of refractory urgency urinary incontinence as compared to the standard injection site protocol (15 injection sites). This endpoint will be measured by reduction in the number of UUI episodes per day.

SECONDARY OUTCOMES:
Quality of life improvement in standard of care (15 injections) versus modified treatment (5 injections) | 6 months
  To compare quality of life and treatment satisfaction scores between the reduced injection site group and the standard injection site group using validated questionnaires. This endpoint will be measured by improvements in numerical scores of patient's perceived quality of life and treatment satisfaction after completion of the procedure.
Complications rates in standard of care (15 injections) versus modified treatment (5 injections) | 6 months
  To determine if the reduced site injection protocol has similar complication rates compared to the standard injection site protocol, specifically: urinary tract infection, post procedure urinary retention, hematuria, pain, and transient weakness. This endpoint will be measured by frequency of complications encountered among each treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Monique J Vaughan, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No